CLINICAL TRIAL: NCT00881296
Title: Randomized Phase II Study of Biweekly Chemotherapy With Gemcitabine and Carboplatin in Elder Patients With Previously Untreated Advanced Non-Small Cell Lung Cancer
Brief Title: Gemcitabine and Carboplatin for Elderly Patient With Lung Cancer
Acronym: GEEP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hamamatsu University (Other)
Responsible Party: Principal Investigator, Naoki Inui, Department of Respiratory Medicine, Hamamatsu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hamamatsu 20-34
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2010-05

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Elder Patients; Non-Small Cell Lung Cancer; Previously Untreated; Advanced
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Gemcitabine 1000mg/m2 Day 1,15
  Carboplatin AUC=3 Day 1, 15 every 4 weeks
  Interventions: Drug: gemcitabine and carboplatin
- 2 (Active Comparator): Gemcitabine 1000mg/m2 Day 1, 8, 15
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: gemcitabine and carboplatin — Gemcitabine 1000mg/m2, DIV on day 1 and 15 of each 28 day cycle. Carboplatin AUC=3, DIV on day 1 and 15 of each 28 day cycle. Number of cycles: until progression or unacceptable toxicity develops, up to 6 cycles.
  Arms: 1
Drug: Gemcitabine — Gemcitabine 1000mg/m2, DIV on day 1, 8 and 15 of each 28 day cycle. Number of cycles: until progression or unacceptable toxicity develops, up to 6 cycles
  Arms: 2

SUMMARY:
A comparison of biweekly combination chemotherapy (gemcitabine plus carboplatin) with weekly gemcitabine in elder patients (> 75) with previously untreated advanced non-small cell lung cancer. Primary objective is to determine the objective response rate (CR+PR by RECIST criteria) for biweekly gemcitabine and carboplatin combination chemotherapy versus weekly single gemcitabine as first-line therapy in elder advanced non-small lung cancer patients (> 76 years) who have received no prior treatment for non-small lung cancer. As secondary objectives, adverse event profile, tolerability of biweekly gemcitabine and carboplatin combination chemotherapy, progression-free survival and overall survival will be evaluated in both patients with biweekly gemcitabine and carboplatin combination chemotherapy and weekly single gemcitabine.

The study hypothesis is that biweekly combination chemotherapy of gemcitabine plus carboplatin may improve the efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed stage IIIB or IV non-small cell lung cancer
* Good performance status (ECOG 0-1)
* No previous treatment
* Age 76 years and older
* Adequate bone marrow, liver and renal functions
* No pregnant
* Measurable disease, defined as at least one lesion whose longest diameter can be accurately measured as >=1.0 cm by spiral CT scan
* Provided written informed consent

Exclusion Criteria:

* Severe complications or a concomitant malignancy
* Prior and other concurrent radiotherapy, chemotherapy, immunotherapy, EGFR tyrosine kinase inhibitors
* Interstitial pneumonia or lung fibrosis
* Contraindicated gemcitabine or carboplatin
* Inappropriate patients for entry to this study, judged by the physicians

Min Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2011-03 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Efficacy (response rate) | two-years, followed RECIST criteria

SECONDARY OUTCOMES:
The toxicity profile (adverse event profile) | two-years, followed NCI-CTCAE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Kingo Chida, MD,PhD, Study Chair — Hamamatsu University
Locations (1):
- Hamamatsu University School of Medicine, Hamamatsu, Shizuoka, Japan

REFERENCES:
- [Derived] Kusagaya H, Inui N, Karayama M, Nakamura Y, Kuroishi S, Yokomura K, Toyoshima M, Shirai T, Masuda M, Yamada T, Yasuda K, Suda T, Chida K. Biweekly combination therapy with gemcitabine and carboplatin compared with gemcitabine monotherapy in elderly patients with advanced non-small-cell lung cancer: a randomized, phase-II study. Lung Cancer. 2012 Sep;77(3):550-5. doi: 10.1016/j.lungcan.2012.05.106. Epub 2012 Jun 15. PMID 22705118